CLINICAL TRIAL: NCT02659930
Title: A Phase 1 Trial of Pomalidomide in Combination With Liposomal Doxorubicin in Patients With Advanced or Refractory Kaposi Sarcoma
Brief Title: Pomalidomide in Combination With Liposomal Doxorubicin in People With Advanced or Refractory Kaposi Sarcoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160047; 16-C-0047
Record Dates: First submitted 2016-01-20; First posted 2016-01-21 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Kaposi Sarcoma
Keywords: HIV; AIDS; Multicentric Castleman Disease
MeSH Terms: conditions — Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Multi-centric Castleman's Disease | interventions — liposomal doxorubicin; pomalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1/Group I (Experimental): Pomalidomide and liposomal doxorubicin given at escalating doses to patients with KS requiring systemic therapy
  Interventions: Drug: liposomal doxorubicin; Drug: pomalidomide
- 2/Group I; Antitumor Assessment Phase (Experimental): Pomalidomide and liposomal doxorubicin, given at the highest tolerated dose to patients with KS requiring systemic therapy
  Interventions: Drug: liposomal doxorubicin; Drug: pomalidomide
- 3/Group II (Experimental): Pomalidomide with liposomal doxorubicin given at escalating doses in to patients with advanced KS or KS and concurrent KSHV-associated MCD or KICS requiring systemic therapy
  Interventions: Drug: liposomal doxorubicin; Drug: pomalidomide
- 4/Group II; Antitumor Assessment Phase (Experimental): Pomalidomide and liposomal doxorubicin, given at the highest tolerated dose to patients with KS or KS with concurrent KSHV-associated MCD or KICS requiring systemic therapy
  Interventions: Drug: liposomal doxorubicin; Drug: pomalidomide

INTERVENTIONS:
Drug: liposomal doxorubicin — liposomal doxorubicin IV day 1 of a 28-day cycle
Drug: pomalidomide — pomalidomide once a day, days 1-21 of a 28-day cycle, at the dose levels described in dose escalation plan

SUMMARY:
Background:

Kaposi sarcoma (KS) is a cancer most often seen in people with HIV. It causes lesions. These are usually on the skin but sometimes in the lymph nodes, lungs, and gastrointestinal tract. Researchers think a combination of drugs may help treat KS.

Objective:

To test a combination of the anti-cancer drugs pomalidomide (CC-4047) and liposomal doxorubicin (Doxil) in people with KS.

Eligibility:

People ages 18 and over with KS

Design:

Participants will be screened with:

Medical history

Questionnaires

Physical exam

Blood, urine, and heart tests

Chest X-ray

Biopsy: A small sample of tissue is taken from a KS lesion.

Possible CT scan

Possible exam of lungs or gastrointestinal tract with an endoscope: A flexible instrument examines

inside the organ.

Participants will take the drugs in 4-week cycles. They will take Doxil through an IV on Day 1 of each cycle. They will take CC-4047 tablets by mouth each day for the first 3 weeks of each cycle.

Participants will have many visits:

Before starting treatment

To start each cycle

Day 15 of first 2 cycles

Visits include repeats of screening tests and:

Multiple blood draws

Photographs of lesions

Participants will keep a drug diary.

Participants will take aspirin or other drugs to prevent blood clots.

Participants with HIV will have combination antiretroviral therapy.

Some participants will have a PET scan.

Participants will continue treatment as long as they tolerate it and their KS improves. After treatment, they will have several follow-up visits for up to 5 years

...

DETAILED DESCRIPTION:
Background:

* Kaposi Sarcoma (KS) is a multicentric angioproliferative tumor that most frequently involves skin, but can also involve lymph nodes, lungs and gastrointestinal tract. It is most common in people with HIV or other forms of immune compromise. Patients with AIDS-associated KS have worse survival than HIV-infected patients without KS.
* Patients may present with advanced disease KS and/or concurrent KSHV-associated multicentric Castleman disease (MCD) or an IL-6 related KSHV-associated cytokine syndrome (KICS). Patients with the latter conditions have poor outcomes when treated with FDA-approved cytotoxic therapies used for KS, and novel approaches are needed.
* A Phase I/II Study demonstrated that pomalidomide 5 mg daily on days 1- 21 of a 28 Day Cycle was safe and tolerable in patients with KS with or without HIV. Increased CD4+ and CD8+ T-cell counts and KS regression were observed.
* Combination of pomalidomide with liposomal doxorubicin may offer a new approach for patients with advanced KS or KS and concurrent KSHV-associated MCD or KICS

Objectives:

* Evaluate the safety and tolerability of various dose combinations of pomalidomide and liposomal doxorubicin in two groups of patients: Group I) KS requiring systemic therapy; Group II) KS with concurrent KSHV-associated MCD or KICS
* To assess the pharmacokinetics (PK) of pomalidomide in combination with liposomal doxorubicin; and for patients with HIV in combination with antiretroviral therapy
* To preliminarily evaluate the antitumor effect of pomalidomide in combination with liposomal doxorubicin against Kaposi sarcoma.

Eligibility:

* Patients with biopsy proven (confirmed in the Laboratory of Pathology, CCR) Kaposi sarcoma (KS)
* Group I: KS requiring systemic therapy (no prior therapy required)

  * T1 KS, KS on skin sufficiently widespread that it is not amenable to local therapy, or KS affecting quality of life due to local symptoms or psychological distress

OR

--KS patients with an inadequate response to pomalidomide (either progressive disease or stable disease after 4 months)

OR

* KS patients with an inadequate response to liposomal doxorubicin, paclitaxel, or other systemic chemotherapy (either progressive disease or stable disease after 6 cycles)
* Group I will exclude patients eligible for Group II (below).
* A wash out period off treatment of 3 weeks will be required, except in the case of patients with progressive, severe disease in which delay of treatment cannot be justified (i.e. symptomatic pulmonary KS)

  -Group II: KS in one of the following high-risk groups (no prior therapy required):
* Concurrent KSHV-associated multicentric Castleman disease (MCD)
* KSHV Inflammatory Cytokine Syndrome (KICS), including those also meeting clinical criteria for KS immune reconstitution syndrome (KS IRIS)

  * Patients with primary effusion lymphoma or a large cell lymphoma arising in KSHV-associated MCD are excluded.

    * At least five measurable cutaneous KS lesions with no previous local radiation, surgical or intralesional cytotoxic therapy that would prevent response assessment for that lesion; or other evaluable disease.
    * ECOG Performance Status (PS): Group I: less than or equal to 2, Group II: less than or equal to 3, ECOG PS of 4 (with Karnofsky 20%) will be allowed in Group II only if symptoms due to pulmonary KS.
    * Measurable disease by the criteria proposed by the AIDS Clinical Trials Group Oncology Committee (for KS).
    * Patient or legal guardian must be willing to give informed consent.
    * Patients can be HIV positive or negative.
    * HAART for HIV+ patients.

Design:

* This is a Phase I study evaluating 2 groups of patients with KS. Patients will receive pomalidomide once a day, days 1-21 of a 28-day cycle, at the various dose levels combined with liposomal doxorubicin IV day 1 of a 28-day cycle until optimal tumor response, unacceptable toxicity, or patient request to discontinue

  * Patients with HIV will be prescribed HAART.
  * All patients will receive thromboprophylaxis, generally with aspirin 81 mg tablet daily.
* The study will proceed to an antitumor activity phase to assess in a preliminary manner the response of Group I patients to a fixed dose of pomalidomide and liposomal doxorubicin. Up to 30 subjects (HIV positive or negative) evaluable for response will be treated at the highest tolerable combination of pomalidomide and liposomal doxorubicin (determined to be dose level 3: pomalidomide 4mg in combination with 20mg/m^2 liposomal doxorubicin) to gain preliminary information on antitumor activity in an expansion cohort. Based on the observation of positive results in the initial dose expansion of 14 patients evaluated in the expansion cohort, a total of 30 patients will be allowed to be included in this cohort in order to gain additional safety information as well as to improve the precision of the estimate of the response rate in Group I patients.
* The study will also include an antitumor activity phase to assess in a preliminary manner the response of Group II patients to a fixed dose of pomalidomide and liposomal doxorubicin. Up to 10 total patients (HIV positive or negative) evaluable for response will be treated at the highest tolerated dose of pomalidomide for this population (determined to be dose level, 2mg in combination with 20mg/m2 liposomal doxorubicin) to gain preliminary information on KS that occurs concurrently with KSHV-MCD or KICS.
* This study will also evaluate the characteristics of 18fluoro-thymidine (FLT) positron emission tomography (PET) in patients with KS and concurrent KSHV-associated MCD or KICS, and correlate with markers of KSHV-lytic activation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed Kaposi sarcoma (KS) confirmed by the Laboratory of Pathology, NCI.
* All patients should have either five measurable cutaneous KS lesions with no previous local radiation, surgical or intralesional cytotoxic therapy that would prevent response assessment for that lesion; or other assessable disease
* Group I: KS requiring systemic therapy (no prior therapy required) and:

  * Group I patients should have one or more of the following:
  * T1 KS, KS on skin sufficiently widespread that it is not amenable to local therapy, or KS affecting quality of life due to local symptoms or psychological distress
  * KS patients with an inadequate response to pomalidomide (either progressive disease or stable disease requiring additional therapy after 4 months)
  * KS patients with an inadequate response to liposomal doxorubicin, paclitaxel, or other systemic chemotherapy (either progressive disease or stable disease requiring additional therapy after 6 cycles)

    * Group I will exclude patients eligible for Group II (below). Patients with a history of multicentric Castleman disease (MCD) in the absence of any active disease (as assessed by the PI) are eligible for Group I.
    * A wash out period off treatment of 3 weeks will be required, except in the case of patients with progressive, severe disease in which delay of treatment cannot be justified (i.e. symptomatic pulmonary KS)
* Group II: KS (no prior therapy required):

  * Concurrent active KSHV-associated multicentric Castleman disease (MCD)
  * Active KSHV Inflammatory Cytokine Syndrome (KICS), including those also meeting clinical criteria for KS immune reconstitution syndrome (KS IRIS)
* At least five measurable cutaneous KS lesions with no previous local radiation, surgical or intralesional cytotoxic therapy that would prevent response assessment for that lesion; or other assessable disease
* ECOG Performance Status (PS):

  * Group I: less than or equal to 2
  * Group II: less than or equal to 3
  * ECOG PS of 4 will be allowed in Group II only if symptoms due to pulmonary KS. (with Karnofsky = 20%).
* Measurable disease by the criteria proposed by the AIDS Clinical Trials Group Oncology Committee (for KS).
* Patients can be HIV positive or negative.
* HAART for HIV+ patients:

  * All HIV+ patients must be willing to be compliant with HAART
  * Group I-on HAART for 1 month with stable disease; however, no minimum time restriction for patients with progressive and/or end-organ threatening disease
  * Group II-no minimum time restriction on prior HAART, patients may be HAART naive.
* Age greater than or equal to 18 years.

  --Because no dosing or adverse event data are currently available on the use of pomalidomide in combination with liposomal doxorubicin in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,000/mcL
  * Platelets >75,000/mcL
  * Hemoglobin

    * Group I: greater than or equal to 8 gm/dL;
    * Group II: if anemia attributed to KS, KSHV-MCD, or KICS greater than or equal to 7gm/dL, otherwise greater than or equal to 8 gm/dL
  * Total bilirubin less than or equal to1.5 upper limit of normal unless the patient is receiving a protease inhibitor known to be associated with increased bilirubin (e.g. atazanavir), in which case total bilirubin less than or equal to 7.5 mg/dL with direct fraction less than or equal to 0.7
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits OR Creatinine clearance >60 mL/min/1.73 m(2) as estimated by either Cockroft-Gault or 24-hour urine collection for patients with creatinine levels above institutional normal
* Cardiac ejection fraction greater than or equal to 50% by echocardiogram
* Patients with a cumulative lifetime history of anthracycline greater than 430 mg/m(2) are eligible, after consultation with a cardiologist, if there are none of the following cardiac risk factors:

  * Diabetes mellitus
  * History of acute coronary syndrome
  * Hypertension; defined as a sustained systolic blood pressure greater than 140 mmHg and/or diastolic blood pressure greater than 90 mmHg OR use of an antihypertensive medication for the indication of hypertension.
* All study participants must agree to be registered into the mandatory POMALYST REMS program, and be willing and able to comply with the requirements of the POMALYST REMS program
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the POMALYST REMSTM program
* Able to take aspirin 81mg daily or if intolerant of aspirin, able to take a substitute thromboprophylaxis such as low molecular weight heparin at a thromboprophylactic dose (such as enoxaparin 0.5mg/kg once daily)
* Because pomalidomide is an agent with the potential for teratogenic or abortifacient effects, females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 14 days prior to and again within 24 hours before starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Patients with primary effusion lymphoma or other concurrent malignancy, except for basal cell carcinoma or squamous carcinoma of the skin or in situ cervical or anal dysplasia
* History of malignant tumors other than KS or KSHV-MCD, unless:

  * In complete remission for greater than or equal to 1 year for the time complete remission was first documented
  * Resected basal cell or squamous cell carcinoma of the skin
  * In situ cervical or anal dysplasia
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of allergic reactions attributed to thalidomide, lenalidomide, or other compounds of similar chemical or biologic composition to pomalidomide or other agents used in study
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pomalidomide, breastfeeding should be discontinued if the mother is treated with pomalidomide. These potential risks may also

apply to other agents used in this study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
safety/tolerability of dose combinations | 3 months
  Incidence of dose limiting toxicity and emerging adverse events
pharmacokinetics of combination therapy | first 3 days of cycle
  Pomalidomide plasma concentrations

SECONDARY OUTCOMES:
Quality of life | 3 months
  assess changes in quality of life in subjects receiving pomalidomide in combination with liposomal doxorubicin
pulmonary function | baseline, cycle 2 and at the end of study
  To assess the effect of the combination on pulmonary function, as measured by pulmonary function tests (PFTs) in patients with pulmonary KS
PET | 3 months
  evaluate the characteristics of 18fluoro-thymidine (FLT) positron emission tomography (PET) in patients with KS and concurrent KSHV-associated MCD or KICS

CONTACTS AND LOCATIONS:
Overall Officials: Ramya M Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@-Genomic data are made available via dbGaP through requests to the data custodians

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0047.html